CLINICAL TRIAL: NCT01912599
Title: Pilot Study on Ambulatory Intraocular Pressure and Blood Pressure Monitoring in Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-2514
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2014-09

CONDITIONS: Normal-Tension Glaucoma
Keywords: Glaucoma; Intraocular Pressure; Blood Pressure
MeSH Terms: conditions — Low Tension Glaucoma; Glaucoma | interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Glaucomatous (Active Comparator): Patients with no history of glaucoma. Subjects will be fitted with Sensimed Triggerfish for 24 observation of IOP and with a blood pressure monitor for 24 hour observation of blood pressure trends.
  Interventions: Device: Sensimed Triggerfish; Device: Blood Pressure
- Glaucoma (Active Comparator): Patients that are currently being treated for moderate to severe normal-tension glaucoma. Subjects will be fitted with Sensimed Triggerfish for 24 observation of IOP and with a blood pressure monitor for 24 hour observation of blood pressure trends.
  Interventions: Device: Sensimed Triggerfish; Device: Blood Pressure

INTERVENTIONS:
Device: Sensimed Triggerfish — IOP will be measured with the Sensimed Triggerfish, which is a disposable silicone contact lens embedded with a wireless sensor. The sensing resistive gauge in the device is circular around the center of the lens and is placed over a circumference of 11.5 mm in diameter. This corresponds to the corneoscleral junction position, where maximum corneal deformation occurs as a result of changes in IOP. A soft patch containing the receiving antenna will be applied around the eye and transmits the information via wire to the recorder that the patient will wear around the waist. The patient can continue to wear spectacles during monitoring. The device records a total of 144 measurements over a 24-hour period.
Device: Blood Pressure — Patients in both groups will be fitted with a blood pressure cuff that will measure pressures for 24 hours.

SUMMARY:
Purpose: To study the feasibility of a larger study by determining the tolerability of measuring blood pressure (BP) and intraocular pressure (IOP) over 24 hours in an ambulatory fashion with automatic devices.

Participants: 20 patients with moderate to severe normal tension glaucoma and 20 non-glaucomatous patients.

Procedures (methods): Both BP and IOP will be measured automatically in each participant in an ambulatory fashion during a 24-hour period. BP will be monitored using an appropriately sized cuff Oscar 2 (Suntech Medical, Morrisville, NC), which will be placed by a person trained in ambulatory BP monitoring devices. The device will be set up to automatically inflate every 30 minutes during the day and every hour during the night to measure and record the BP. IOP will be measured using Sensimed Triggerfish contact lens (Sensimed AG, Lausanne, Switzerland); the measurements will be taken and recorded every 10 minutes. The contact lens will be inserted by eye doctors (investigators). Both monitoring devices will be removed the following day.

DETAILED DESCRIPTION:
Chart review will be performed to select potential glaucoma participants. These potential participants will be invited to participate in the study, either by phone or face-to-face during scheduled visits.

Control participants will be invited from a registry that contains names of prior research participants who have agreed to be contacted about future studies (participants have worn ambulatory blood pressure monitor or ABPM in the past).

Invited persons who agree to participate in the study will be scheduled for a screening visit at the eye clinic, during which they will learn more about the study. On the day of the screening visit, they will be provided with detailed information about the study, after which they will decide whether or not to participate. If they agree, they will sign the consent form. The screening visit will then be conducted by the research personnel and will take place at the eye clinic in a designated closed office and will include measurement of visual acuity, assessment of the anterior and posterior segments of the eye, measurement of IOP by Goldmann applanation tonometry. If after the screening exam it is determined that they do not qualify for the study, they will be told why they are being excluded. Healthy controls as well as glaucomatous patients not on treatment will be fitted with the BP and IOP monitoring devices. Those who are on glaucoma medication will be asked to stop their medication starting the day following the screening visit for the duration detailed in the inclusion criteria, and be given an appointment for the for IOP and BP measurement. On the appointment day, they will be fitted the BP and IOP monitoring devices. The BP monitor will be set up to take the measurements automatically every 30 min during the day and every hour at night until the next morning. The IOP monitor will take measurements every 10 minutes during the 24-hour period. Both devices are computerized and record all the measurements and reading times. Patients will be required to return to the clinic the next morning for removal of the devices, after which there will be no further visits.

1. This study will provide for the first time information on the safety, tolerance, and acceptability of the two devices used together. It will also provide preliminary information on the reasons why people may drop out of the study, and information about the relationship between IOP, BP, and OPP in patients with normal tension glaucoma and in healthy controls.
2. IOP will be measured with the Sensimed Triggerfish, which is a disposable silicone contact lens embedded with a wireless sensor. The sensing resistive gauge in the device is circular around the center of the lens and is placed over a circumference of 11.5 mm in diameter. This corresponds to the corneoscleral junction position, where maximum corneal deformation occurs as a result of changes in IOP. A soft patch containing the receiving antenna will be applied around the eye and transmits the information via wire to the recorder that the patient will wear around the waist. The patient can continue to wear spectacles during monitoring. The device records a total of 144 measurements over a 24-hour period. Measurements are taken every 10 min for a total duration of 1 min. The results obtained are presented in an arbitrary unit and not mm Hg. In this study, tonometry will be performed using radiofrequency waves at 27 MHz from the external antenna, which is embedded in the patch applied around the patient's eye.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with normal tension glaucoma

  * Age minimum: 18 years
  * Willingness to participate in the study and to sign the informed consent form.
  * Willingness to complete a screening visit and a study visit, both at the UNC eye clinic.
  * Established diagnosis of untreated or medically treated normal tension glaucoma irrespective of blood pressure level. Those currently treated with topical drops will only be included in the study if they accept to stop their medication according to the following plan: 1) Those treated with Alphagan, Combigan or Cosopt (or Trusopt, Azopt, Diamox, Neptazane) will be asked to stop their medication for a week, do the study for 24 hours, and then resume with their medication. 2) Those treated with Timolol or Xalatan (or Travatan, Lumigan) will be asked to stop their drops for one month, do the study for 24 hours, and then resume the medication regimen. The reason for this is that the study aims at investigating the relationship between blood pressure and intraocular pressure in untreated patients either for glaucoma or high blood pressure. The difference in duration of time during which patients will be off their glaucoma medication depends on the time it takes to clear the drug in the system. In both cases, glaucoma medication will be stopped from the day following the screening visit.

    2) Non-glaucomatous healthy controls
  * Age minimum: 18 years
  * Willingness to participate in the study and to sign a consent form
  * Willingness to complete a screening visit at UNC eye clinic
  * Normal eye examination

Exclusion Criteria:

* 1) Patients with normal tension glaucoma

  * Age less than 18 years or greater than 80 years.
  * Patients with high intraocular pressure (> 21 mmHg).
  * Patients who have had any type of glaucoma surgery in the past.
  * Non-glaucomatous optic neuropathy.
  * Intraocular surgery within the last 3 months.
  * Patients with uveitis
  * Ocular abnormalities preventing measurement of intraocular pressure by applanation
  * Patients on medication to treat high blood pressure will not be included in the study.
  * Patients with hyperthyroidism
  * Patients on medication that may raise blood pressure: i.e. systemic or topical steroids taken for 3 or more years for other chronic conditions; cholesterol lowering medications, specifically cholestyramine (Prevalite or Questran) or colestipol (Colestid); oral contraceptives that contain higher concentrations of estrogen, specifically: Ovral, Ogestrel, Demulen, Ovon, and Ortho-Novum; and the antidepressants trimipramine (Surmontil) and venlafaxine (Effexor).
  * Patients on estrogen taken for menopause because it may lower blood pressure
  * Patients not willing to stop their glaucoma medication temporarily
  * Patients with dry eye disease

    2) Control Patients
    * Age less than 18 years or greater than 80 years.

      * Patients with high intraocular pressure (> 21 mmHg).
      * Patients who have had any type of glaucoma surgery in the past.
      * Non-glaucomatous optic neuropathy.
      * Intraocular surgery within the last 3 months.
      * Patients with uveitis
      * Ocular abnormalities preventing measurement of intraocular pressure by applanation
      * Patients on medication to treat high blood pressure will not be included in the study.
      * Patients with hyperthyroidism
      * Patients on medication that may raise blood pressure: i.e. systemic or topical steroids taken for 3 or more years for other chronic conditions; cholesterol lowering medications, specifically cholestyramine (Prevalite or Questran) or colestipol (Colestid); oral contraceptives that contain higher concentrations of estrogen, specifically: Ovral, Ogestrel, Demulen, Ovon, and Ortho-Novum; and the antidepressants trimipramine (Surmontil) and venlafaxine (Effexor).
      * Patients on estrogen taken for menopause because it may lower blood pressure
      * Patients with dry eye disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Mwanza, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Kittner Eye Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Glaucomatous | Glaucoma
Started | 20 | 16
Completed | 20 | 15
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: N/A Pilot Study
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Glaucomatous | Glaucoma | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 8 | 26
  >=65 years | 2 | 8 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (13.3) | 66.9 (11.1) | 57.3 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 13 | 7 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Arterial Pressure
Description: The blood pressure value shown in the table is the mean of all measurements taken over the 24 hour period, so it is the average value.
Time Frame: 24 Hours
Population: Data for two glaucoma patients were excluded for analysis because
  * In one patient the IOP recorder malfunctioned just two hours after set up, so data were not available for the entire 24 hours
  * In the other patient, the wireless sensor was disconnected from the recorder in the middle if the night so data could not be recorded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Non-Glaucomatous | Glaucoma
Number analyzed (Participants) | 20 | 13
mmHg | 100.9 (23.6) | 95.5 (11.4)

2. Primary Outcome: Intraocular Pressure
Description: The IOP provided is the average of all 144 measurements taken during the 24 hour period.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: mEqv.
Arm/Group | Non-Glaucomatous | Glaucoma
Number analyzed (Participants) | 20 | 15
mEqv. | 17.6 (126.5) | 179.2 (87.2)

3. Primary Outcome: Mean Perfusion Pressure
Description: The value shown in the table is the mean of all measurements taken over the 24 hour period, so it is the average value.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Non-Glaucomatous | Glaucoma
Number analyzed (Participants) | 20 | 15
mmHg | 90.8 (135.6) | 62.4 (12.7)

4. Primary Outcome: Diastolic Pressure
Description: The value shown in the table is the mean of all measurements taken over the 24 hour period, so it is the average value.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Non-Glaucomatous | Glaucoma
Number analyzed (Participants) | 20 | 15
mmHg | 85.7 (9.3) | 74.6 (11.6)

5. Primary Outcome: Systolic Pressure
Description: The value shown in the table is the mean of all measurements taken over the 24 hour period, so it is the average value.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Non-Glaucomatous | Glaucoma
Number analyzed (Participants) | 20 | 15
mmHg | 146.4 (15.2) | 129.0 (35.2)

ADVERSE EVENTS:
Arm/Group | Non-Glaucomatous | Glaucoma
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 7/20 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Glaucomatous (N=20) | Glaucoma (N=16)
Corneal Changes (Eye disorders) | 6 (6) | 3 (3) — Includes Epithelial Disruption, corneal edema, and Descemet's folds.
Conjunctival Changes (Eye disorders) | 1 (1) | 3 (3) — Chemosis and conjunctival disruption.
Cuff Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Arm had an abrasion due to blood pressure cuff.

LIMITATIONS AND CAVEATS:
The limitation is that the contact lens expresses the IOP values in a unit that is not convertible to mmHg. Therefore, we do not know exactly what the cutoff of normal IOP with the lens is.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No